CLINICAL TRIAL: NCT03232801
Title: A Mindfulness-based Intervention for Older Women With Low Sexual Desire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Holly Thomas, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRO15060240; K23AG052628 (NIH)
Record Dates: First submitted 2017-03-10; First posted 2017-07-28 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Hypoactive Sexual Desire Disorder; Sexual Dysfunction; Female Sexual Dysfunction
Keywords: hypoactive sexual desire disorder; female sexual dysfunction; low libido; female sexual interest-arousal disorder; low desire; sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness group (Experimental): A multicomponent group-based intervention rooted in mindfulness, administered in 3 sessions over 6 weeks
  Interventions: Behavioral: mindfulness-based multicomponent intervention
- educational group (Active Comparator): A general midlife health and aging educational group, administered in 3 sessions over 6 weeks
  Interventions: Behavioral: general health education group

INTERVENTIONS:
Behavioral: mindfulness-based multicomponent intervention — A group-based, multicomponent behavioral intervention rooted in mindfulness
  Arms: mindfulness group
Behavioral: general health education group — A general health and aging education group
  Arms: educational group

SUMMARY:
The overall aim of this research is to adapt and pilot test a multi-component, mindfulness-based behavioral intervention for women age 50 and older with low sexual desire.

DETAILED DESCRIPTION:
Specifically, the investigators will conduct a pilot randomized controlled trial to assess the feasibility, acceptability, and preliminary efficacy of the intervention. Fifty women will be randomized to the mindfulness intervention or an educational control group. Both groups will be conducted in 3 sessions over 6 weeks in groups of 10 women. Feasibility, acceptability, facilitators, and barriers will be assessed by surveys after each session and after intervention completion. Preliminary efficacy will be assessed by measures of sexual desire, sexual function, and overall sexual satisfaction at 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for a diagnosis of Female Sexual Interest/Arousal Disorder
* English-speaking
* have a current sexual partner with whom they are or would like to be sexually active

Exclusion Criteria:

* active major depression
* active substance abuse
* current intimate partner violence
* partner with active major depression
* partner with active major substance abuse
* significant relationship dissatisfaction
* current use of antidepressants
* untreated dyspareunia (sexual pain)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women participants only
Enrollment: 62 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 women were screened. 19 women were ineligible (N=62 enrolled). One woman withdrew after consent but before randomization. N=61 women were randomized.
Period: Overall Study
Arm/Group | Mindfulness Group | Educational Group
Started | 31 | 30
Completed Baseline Survey | 28 | 27
Attended at Least One Session | 18 | 23
Completed Week 7 Follow-up | 15 | 22
Completed Week 12 Follow-up | 15 | 18
Completed | 15 | 18
Not Completed | 16 | 12

BASELINE CHARACTERISTICS:
Population: 61 participants were randomized, but only 55 participants completed baseline assessments
Groups:
- Mindfulness: A six-session mindfulness-based intervention focused on sexual health and function. Groups met weekly for 1.5-2 hours over the course of six weeks. Groups were co-led by a primary care physician (the primary investigator) and a trained mindfulness instructor with over 10 years of experience in mindfulness meditation instruction. The intervention contained elements of mindfulness-based stress reduction and sexual psychoeducation. Intervention components including instruction in mindfulness meditation, body scan, awareness of breathing, mindful yoga, and loving kindness meditation, as well as application of these practices to sexual function. At least 30 minutes of each session were spent in mindfulness practice. Sessions also included group discussions and break-out rooms to facilitate discussinos about the practice. Based on prior qualitative research, the intervention also included information about partner sexual dysfunction, body image, and how menopause can affect sexuality. Participants were encouraged to do 60 minutes of mindfulness home practice daily and were provided with audio recordings to facilitate home practice. Home practice included sexuality-specific mindfulness exercises.
- Education: The control condition was a six-session health education intervention. Groups met weekly for 1.5-2 hours over the course of six weeks. Groups were led by a primary care physician (the primary investigator) alone. The control intervention covered general educational topics relevant to the health of midlife women, such as osteoporosis and heart disease. Sexual health was discussed in one session, but not in detail. At the conclusion of their participation in the group, control group participants were given a brochure with local resources for learning about mindfulness meditation. Participants did not have any homework to complete for this group.
- Total: Total of all reporting groups
Arm/Group | Mindfulness | Education | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (7.1) | 55.7 (7.5) | 55.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 20 | 24 | 44
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55
Female Sexual Function Index (FSFI) [Mean (Standard Deviation); unit: units on a scale] — The Female Sexual Function Index (FSFI) is a 19-item self-report inventory designed to assess female sexual function. It comprises six domains: desire [two items], arousal [four items], lubrication [four items], orgasm, satisfaction, pain [three items each]. The FSFI total score is the sum of the 6 domain/subscale scores. The minimum score is 2.0. The maximum score is 36.0. Higher scores indicate worse functioning. A total score 26.0 has been validated as a cutoff score for diagnosing Female Sexual Dysfunction.
  units on a scale | 21.1 (6.1) | 20.5 (7.3) | 20.7 (6.7)
Female Sexual Distress Scale - Revised (FSDS-R) [Mean (Standard Deviation); unit: units on a scale] — The Female Sexual Distress Scale-Revised (FSDS-R) was created and validated to assess distress associated with impaired sexual function. It contains 13 items. The total score, ranging from 0 to 48, provides a measure of sexual distress, in which the higher the score, the higher the level of sexual distress.
  units on a scale | 23.3 (11.9) | 18.5 (8.8) | 20.7 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Number of Enrolled Women Participating in All Sessions
Description: Number of enrolled women participating in all sessions
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Mindfulness: Assigned to mindfulness-based intervention group
- Education: Assigned to general menopause education group
Arm/Group | Mindfulness | Education
Number analyzed (Participants) | 31 | 30
Participants | 15 | 22
Statistical Analysis 1: Comparison: Mindfulness vs Education; Test type: Superiority; p = 0.027, Chi-squared; chi-squared = 4.86

2. Primary Outcome: Acceptability - Number of Women Indicating "Somewhat" or "Very Satisfied" on a 5-point Likert Scale Measure of Intervention Satisfaction
Description: Number of women indicating "somewhat" or "very satisfied" on a 5-point Likert scale measure of intervention satisfaction
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Group | Educational Group
Number analyzed (Participants) | 15 | 22
Participants | 14 | 19
Statistical Analysis 1: Comparison: Mindfulness Group vs Educational Group; Test type: Superiority; p = 0.503, Chi-squared; chi-squared = 0.45

3. Secondary Outcome: Change in FSFI Desire Score
Description: Change in Female Sexual Function Index (FSFI) desire score from baseline to 12 weeks. The FSFI Desire score is a subscale of the FSFI. Scores range from 1.0 to 5.0, with higher scores indicating worse sexual desire. Minimum score is 1.0 and maximum score is 5.0.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness | Education
Number analyzed (Participants) | 15 | 18
units on a scale | 0.4 (0.8) | 0.7 (0.7)

4. Other Pre Specified Outcome: Change in Overall Sexual Function
Description: Total Female Sexual Function Index (FSFI) score from baseline to 12 weeks. The FSFI score can range from 2.0 to 36.0, and a higher score indicates worse sexual function.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness | Education
Number analyzed (Participants) | 15 | 18
units on a scale | 4.0 (5.1) | 1.5 (3.0)

5. Other Pre Specified Outcome: Comprehensive Sexual Desire
Description: Sexual Interest and Desire Inventory (SIDI)
Time Frame: 6 weeks and 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Sexual Distress
Description: Female Sexual Distress Scale - Revised (FSDS-R)
Time Frame: 6 weeks and 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Quality of Life - SF 36
Description: Quality of life as measured by Short Form-36 (SF-36)
Time Frame: 6 weeks and 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Mindfulness Group | Educational Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03232801/Prot_001.pdf
  • Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03232801/SAP_002.pdf